CLINICAL TRIAL: NCT02486406
Title: An Open-Label, Multicenter Study to Evaluate the Pharmacokinetics, Safety, and Efficacy of Ombitasvir (OBV), Paritaprevir (PTV), Ritonavir (RTV) With or Without Dasabuvir (DSV) and With or Without Ribavirin (RBV) in Pediatric Subjects With Genotype 1 or 4 Chronic Hepatitis C Virus (HCV) Infection (ZIRCON)
Brief Title: A Study to Evaluate Treatment of Hepatitis C Virus Infection in Pediatric Subjects
Acronym: ZIRCON
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-748; 2015-000111-41 (EudraCT Number)
Record Dates: First submitted 2015-06-17; First posted 2015-07-01 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C Virus; Hepatitis C Genotype 1; Hepatitis C Genotype 4; Pediatric
MeSH Terms: conditions — Hepatitis C | interventions — ombitasvir; paritaprevir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Adult tablet, 12-17 yr, Part 1 (Experimental): Participants with HCV GT1b without cirrhosis received the adult 3-DAA (OBV/PTV/RTV and DSV) regimen: two 12.5 mg ombitasvir /75 mg paritaprevir /50 mg ritonavir tablets taken orally every morning (QD) and one dasabuvir 250 mg tablet taken orally twice a day (BID) for 12 weeks. Participants with HCV GT1a without cirrhosis received 12-week treatment with the adult 3-DAA regimen and ribavirin 200 mg tablets were administered orally per local label.
  Interventions: Drug: Ombitasvir/paritaprevir/ritonavir; Drug: Dasabuvir; Drug: Ribavirin
- Adult tablet, 12-17 yr, Part 2 (Experimental): Participants with HCV GT1b received the adult 3-DAA (OBV/PTV/RTV and DSV) regimen: two 12.5 mg ombitasvir /75mg paritaprevir /50 mg ritonavir tablets taken orally every morning (QD) and one dasabuvir 250 mg tablet taken orally twice a day (BID) for 12 weeks. Participants with HCV GT1a without cirrhosis received 12-week treatment with the adult 3-DAA regimen and ribavirin 200 mg tablets were administered orally per local label. Participants with HCV GT1a with compensated cirrhosis received 24-week treatment with the adult 3-DAA regimen and ribavirin 200 mg tablets were administered orally per local label. Participants with HCV GT4 received 12-week treatment with the OBV/PTV/RTV formulation and ribavirin 200 mg tablets were administered orally per local label.
  Interventions: Drug: Ombitasvir/paritaprevir/ritonavir; Drug: Dasabuvir; Drug: Ribavirin
- Mini tablet, 9-11 yr, Part 1 (Experimental): Participants with HCV GT1b without cirrhosis were to receive the mini-tablet 3-DAA (OBV, PTV, RTV, and DSV) regimen for 12 weeks: ombitasvir 0.3 mg, paritaprevir 1.0 mg, and ritonavir 1.0 mg mini-tablets administered orally QD based on body weight and dasabuvir taken orally BID as 3.08 mg mini-tablets based on body weight. Participants with HCV GT1a without cirrhosis received 12-week treatment with the mini-tablet 3-DAA regimen and ribavirin was provided as a 40 mg/mL oral solution and administered per local label.
  Interventions: Drug: Ombitasvir mini tablet; Drug: Paritaprevir mini tablet; Drug: Ritonavir mini tablet; Drug: Dasabuvir mini tablet; Drug: Ribavirin solution
- Mini tablet, 3-8 yr, Part 1 (Experimental): Participants with HCV GT1b without cirrhosis were to receive the mini-tablet 3-DAA (OBV, PTV, RTV, and DSV) regimen for 12 weeks: ombitasvir 0.3 mg, paritaprevir 1.0 mg, and ritonavir 1.0 mg mini-tablets administered orally QD based on body weight and dasabuvir taken orally BID as 3.08 mg mini-tablets based on body weight. Participants with HCV GT1a without cirrhosis received 12-week treatment with the mini-tablet 3-DAA regimen and ribavirin was provided as a 40 mg/mL oral solution and administered per local label.
  Interventions: Drug: Ombitasvir mini tablet; Drug: Paritaprevir mini tablet; Drug: Ritonavir mini tablet; Drug: Dasabuvir mini tablet; Drug: Ribavirin solution

INTERVENTIONS:
Drug: Ombitasvir/paritaprevir/ritonavir — Film-coated tablet for oral use
  Other Names: Ombitasvir also known as ABT-267; Paritaprevir also known as ABT-450; Ombitsvir/paritaprevir/ritonavir also known as Viekirax
  Arms: Adult tablet, 12-17 yr, Part 1; Adult tablet, 12-17 yr, Part 2
Drug: Dasabuvir — Film-coated tablet for oral use
  Other Names: Exviera; ABT-333
  Arms: Adult tablet, 12-17 yr, Part 1; Adult tablet, 12-17 yr, Part 2
Drug: Ribavirin — Film-coated tablet for oral use
  Arms: Adult tablet, 12-17 yr, Part 1; Adult tablet, 12-17 yr, Part 2
Drug: Ombitasvir mini tablet — Film-coated tablet for oral use
  Other Names: ABT-267
  Arms: Mini tablet, 3-8 yr, Part 1; Mini tablet, 9-11 yr, Part 1
Drug: Paritaprevir mini tablet — Film-coated tablet for oral use
  Other Names: ABT-450
  Arms: Mini tablet, 3-8 yr, Part 1; Mini tablet, 9-11 yr, Part 1
Drug: Ritonavir mini tablet — Film-coated tablet for oral use
  Arms: Mini tablet, 3-8 yr, Part 1; Mini tablet, 9-11 yr, Part 1
Drug: Dasabuvir mini tablet — Film-coated tablet for oral use
  Other Names: Exviera; ABT-333
  Arms: Mini tablet, 3-8 yr, Part 1; Mini tablet, 9-11 yr, Part 1
Drug: Ribavirin solution — Oral solution
  Arms: Mini tablet, 3-8 yr, Part 1; Mini tablet, 9-11 yr, Part 1

SUMMARY:
This was a Phase 2/3, open-label, multicenter study to evaluate the pharmacokinetics (PK), efficacy, and safety of ombitasvir/paritaprevir/ritonavir (OBV/PTV/RTV) with or without dasabuvir (DSV) and with or without ribavirin (RBV) in Hepatitis C virus (HCV) genotype 1 or 4 (GT1 or GT4)-infected pediatric participants of ≥ 3 to 17 years of age.

DETAILED DESCRIPTION:
The study population for Part 1, the PK study, included GT1-infected participants who were noncirrhotic and treatment-naïve (TN). Part 2, the safety and efficacy study, included GT1 or GT4-infected participants who were TN or interferon ([IFN] or Pegylated-interferon alfa-2a or 2b [pegIFN] with or without RBV) treatment-experienced (TE) without cirrhosis or with compensated cirrhosis. In Part 1 and Part 2, the treatment regimen and duration were dependent on HCV GT, GT1 subtype, and cirrhosis status.

ELIGIBILITY:
Inclusion Criteria:

1. Positive anti-hepatitis C virus antibody (HCV Ab) and HCV ribonucleic acid (RNA) ≥ 1000 IU/mL at the time of screening
2. HCV genotype 1 for enrollment into Part 1 of the study and genotype 1 or 4 for enrollment into Part 2
3. Parent or legal guardian with the willingness and ability to provide written informed consent and participant willing and able to give assent, as appropriate for age and country

Exclusion Criteria:

1. Female participant who is pregnant, breastfeeding or is considering becoming pregnant
2. Use of known strong inducers and inhibitors (e.g., gemfibrozil) of cytochrome P450 2C8 (CYP2C8) in participants receiving dasabuvir, or strong or moderate inducers of CYP3A, within 2 weeks or 10 half-lives, whichever is longer, of the respective medication/supplement prior to study drug administration.
3. Positive test result for Hepatitis B surface antigen (HbsAg) or anti-human immunodeficiency virus antibody (HIV Ab) test
4. Current enrollment in another interventional clinical study, previous enrollment in this study, prior or current use of any investigational or commercially available anti-HCV agents other than interferons or ribavirin or receipt of any investigational product within 6 weeks prior to study drug administration

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (21):
- United States (11):
  - UCSF Benioff Childrens Hosp /ID# 136774, San Francisco, California
  - Children's Hospital Colorado /ID# 137017, Aurora, Colorado
  - University of Florida - Archer /ID# 136830, Gainesville, Florida
  - Advent Health /ID# 167663, Orlando, Florida
  - Indiana University /ID# 137015, Indianapolis, Indiana
  - Boston Childrens Hospital /ID# 137174, Boston, Massachusetts
  - Boston Medical Center /ID# 136831, Boston, Massachusetts
  - Columbia Univ Medical Center /ID# 136431, New York, New York
  - Children's Hospital of Philadelphia /ID# 137018, Philadelphia, Pennsylvania
  - Baylor College of Medicine /ID# 136590, Houston, Texas
  - Seattle Children's Hospital /ID# 137019, Seattle, Washington
- Belgium (2):
  - Cliniques Universitaires Saint-Luc /ID# 136910, Brussels, Brussels Capital
  - UZ Leuven /ID# 136911, Leuven
- Germany (3):
  - Charite Universitaetsmedizin Berlin /ID# 141620, Berlin
  - Universitaetsklinikum Freiburg /ID# 141618, Freiburg im Breisgau
  - Helios Klinikum Wuppertal /ID# 142883, Wuppertal
- San Jorge Children Hospital /ID# 136832, San Juan, Puerto Rico
- Spain (4):
  - Hospital Sant Joan de Deu /ID# 137096, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 137098, Barcelona
  - Hospital Universitario La Paz /ID# 137094, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 137097, Valencia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Rosenthal P, Narkewicz MR, Yao BB, Jolley CD, Lobritto SJ, Wen J, Molleston JP, Hsu EK, Jonas MM, Zha J, Liu L, Leung DH. Ombitasvir, Paritaprevir, Ritonavir, and Dasabuvir Mini-Tabs Plus Ribavirin for Children Aged 3-11 Years with Hepatitis C Genotype 1a. Adv Ther. 2020 Jul;37(7):3299-3310. doi: 10.1007/s12325-020-01389-9. Epub 2020 May 25. PMID 32451952

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety population: all participants who received at least one dose of study drug in Part 1 or Part 2
Period: Overall Study
Arm/Group | Adult Tablet, 12-17 yr, Part 1 | Adult Tablet, 12-17 yr, Part 2 | Mini Tablet, 9-11 yr, Part 1 | Mini Tablet, 3-8 yr, Part 1
Started | 12 | 26 | 12 | 14
Completed | 10 | 23 | 10 | 10
Not Completed | 2 | 3 | 2 | 4
Not completed — Withdrew consent | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 3 | 1 | 3
Not completed — Other, not specified | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population: all participants who received at least one dose of study drug in Part 1 or Part 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult Tablet, 12-17 yr, Part 1 | Adult Tablet, 12-17 yr, Part 2 | Mini Tablet, 9-11 yr, Part 1 | Mini Tablet, 3-8 yr, Part 1 | Total
Number analyzed (Participants) | 12 | 26 | 12 | 14 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.73) | 15.0 (1.68) | 9.8 (0.83) | 4.8 (1.67) | 11.9 (4.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 6 | 11 | 42
  Male | 3 | 10 | 6 | 3 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 23 | 10 | 10 | 49
  Black or African American | 2 | 3 | 0 | 4 | 9
  Asian | 3 | 0 | 1 | 0 | 4
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Multi race | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of Ombitasvir (OBV)
Description: Cmax is the peak concentration that a drug or drug metabolite achieves in a specified compartment after the drug has been administrated and before administration of a second dose.
Time Frame: At Week 2
Population: Intention-to-treat population: all participants who received at least one dose of study drug in Part 1 with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 15 - 29 kg Body Weight: Participants in Part 1 of the study who weighed between 15-29 kg at the time of enrollment
- 30 - 44 kg Body Weight: Participants in Part 1 of the study who weighed between 30-44 kg at the time of enrollment
- ≥ 45 kg Body Weight: Participants in Part 1 of the study who weighed ≥ 45 kg at the time of enrollment
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 9 | 13
ng/mL | 99.6 (27) | 116 (14) | 83.7 (39)

2. Primary Outcome: Part 1: Concentration of Drug in Blood Plasma Over Time [Area Under the Curve (AUC)] of Ombitasvir (OBV)
Description: AUC is a measure of how long and how much drug is present in the body after dosing. The amount of ombitasvir present was measured up to 24 hours after dosing.
Time Frame: At Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 8 | 12
ng•h/mL | 1270 (26) | 1490 (12) | 1060 (43)

3. Primary Outcome: Part 1: Lowest Plasma Concentration (Ctrough) of Ombitasvir (OBV)
Description: Minimum plasma concentration (Ctrough; measured in ng/mL) was directly determined from the concentration-time data.
Time Frame: At Weeks 2 and 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 8 | 12
ng/mL
  Week 2 | 24.7 (32) | 28.2 (16) | 21.8 (39)
  Week 8: number analyzed (Participants) | 11 | 7 | 11
  Week 8 | 29.6 (78) | 30.4 (24) | 20.9 (58)

4. Primary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of Paritaprevir (PTV)
Description: as for outcome 1
Time Frame: At Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 9 | 13
ng/mL | 294 (152) | 1540 (71) | 870 (125)

5. Primary Outcome: Part 1: Concentration of Drug in Blood Plasma Over Time [Area Under the Curve (AUC)] of Paritaprevir (PTV)
Description: AUC is a measure of how long and how much drug is present in the body after dosing. The amount of paritaprevir present was measured up to 24 hours after dosing.
Time Frame: At Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 8 | 12
ng•h/mL | 2180 (136) | 8640 (90) | 5770 (152)

6. Primary Outcome: Part 1: Lowest Plasma Concentration (Ctrough) of Paritaprevir (PTV)
Description: Minimum plasma concentration (Ctrough; measured in ng/mL) was directly determined from the concentration-time data.
Time Frame: At Weeks 2 and 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 8 | 12
ng/mL
  Week 2 | 9.86 (113) | 16.1 (112) | 18.0 (78)
  Week 8: number analyzed (Participants) | 12 | 7 | 11
  Week 8 | 17.3 (136) | 18.4 (89) | 23.5 (86)

7. Primary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of Dasabuvir (DSV)
Description: as for outcome 1
Time Frame: At Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 9 | 13
ng/mL | 579 (44) | 830 (45) | 671 (48)

8. Primary Outcome: Part 1: Concentration of Drug in Blood Plasma Against Time [Area Under the Curve (AUC)] of Dasabuvir (DSV)
Description: AUC is a measure of how long and how much drug is present in the body after dosing. The amount of dasabuvir present was measured up to 12 hours after dosing. For two subjects in the 15-29 kg group, the 24 h concentration was used as the 12 h concentration due to the significant sampling time deviation. For one subject in the 30-44 kg group, the 24 h concentration was used as the 12 h concentration due to the significant sampling time deviation.
Time Frame: At Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 9 | 13
ng•h/mL | 3960 (44) | 5960 (47) | 4630 (49)

9. Primary Outcome: Part 1: Lowest Plasma Concentration (Ctrough) of Dasabuvir (DSV)
Description: Minimum plasma concentration (Ctrough; measured in ng/mL) was directly determined from the concentration-time data.
Time Frame: At Weeks 2 and 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 9 | 13
ng/mL
  Week 2 | 110 (57) | 215 (54) | 165 (56)
  Week 8: number analyzed (Participants) | 12 | 7 | 11
  Week 8 | 168 (82) | 264 (65) | 191 (60)

10. Primary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of Ritonavir (RTV)
Description: as for outcome 1
Time Frame: At Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 9 | 13
ng/mL | 1090 (67) | 1830 (42) | 1180 (35)

11. Primary Outcome: Part 1: Concentration of Drug in Blood Plasma Over Time [Area Under the Curve (AUC)] of Ritonavir (RTV)
Description: AUC is a measure of how long and how much drug is present in the body after dosing. The amount of ritonavir present was measured up to 24 hours after dosing.
Time Frame: At Week 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 9 | 12
ng•h/mL | 6570 (60) | 14100 (49) | 8900 (37)

12. Primary Outcome: Part 1: Lowest Plasma Concentration (Ctrough) of Ritonavir (RTV)
Description: Minimum plasma concentration (Ctrough; measured in ng/mL) was directly determined from the concentration-time data.
Time Frame: At Weeks 2 and 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 15 - 29 kg Body Weight | 30 - 44 kg Body Weight | ≥ 45 kg Body Weight
Number analyzed (Participants) | 12 | 9 | 12
ng/mL
  Week 2 | 16.1 (72) | 32.1 (63) | 29.8 (54)
  Week 8: number analyzed (Participants) | 12 | 7 | 11
  Week 8 | 91.8 (268) | 38.1 (112) | 58.2 (138)

13. Primary Outcome: Parts 1 and 2: Percentage of Participants With Sustained Virologic Response 12 Weeks After the Last Actual Dose of Study Drug (SVR12)
Description: SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) < lower limit of quantification (LLOQ) 12 weeks after the last actual dose of study drug.
Time Frame: 12 weeks after last dose of study drug (Week 24 or 36 depending on treatment duration)
Population: Intention-to-treat population: all participants who received at least one dose of study drug in Part 1 or 2; those with missing data after backwards imputation were treated as nonresponders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants, Total: All participants who received at least one dose of study drug in Part 1 or Part 2
Arm/Group | All Participants, Total
Number analyzed (Participants) | 64
percentage of participants | 98.4 [91.7 to 99.7]
Statistical Analysis 1: Comparison: All Participants, Total; According to the Highlights of Prescribing Information of PEGASYS, the SVR24 rate was 47% among 45 treatment-naïve pediatric participants with HCV GT1 in the NV17424 trial. To show that the DAA regimen is superior to this current standard of care by 20%, the lower bound of the 2-sided 95% confidence interval of the SVR12 rate across all participants in the study must be greater than 67%; Test type: Superiority; Wilson's score method = 98.4, 95% CI 2-sided [91.7 to 99.7]

14. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Sustained Virologic Response 12 Weeks After the Last Actual Dose of Study Drug (SVR12) Summarized by Formulation, Age and Weight Group, and Across All Subjects on the Adult Formulations
Description: as for outcome 13
Time Frame: 12 weeks after last dose of study drug (Week 24 or 36 depending on treatment duration)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Adult Tablet, 12-17 YR, ≥ 45 kg: Participants age 12-17 years old who received the adult formulation and weighed ≥ 45 kg
- Mini-tablet, 9-11 YR, 15 to 29 kg: Participants age 9-11 years old who received the mini-tablet formulation and weighed 15 to 29 kg
- Mini-tablet, 9-11 YR, 30 to 44 kg: Participants age 9-11 years old who received the mini-tablet formulation and weighed 30 to 44 kg
- Mini-tablet, 9-11 YR, ≥ 45 kg: Participants age 9-11 years old who received the mini-tablet formulation and weighed ≥ 45 kg
- Mini-tablet, 3-8 YR, 15 to 29 kg: Participants age 3-8 years old who received the mini-tablet formulation and weighed 15 to 29 kg
- Mini-tablet Total: All participants who received the mini-tablet formulation
Arm/Group | Adult Tablet, 12-17 YR, ≥ 45 kg | Mini-tablet, 9-11 YR, 15 to 29 kg | Mini-tablet, 9-11 YR, 30 to 44 kg | Mini-tablet, 9-11 YR, ≥ 45 kg | Mini-tablet, 3-8 YR, 15 to 29 kg | Mini-tablet Total
Number analyzed (Participants) | 38 | 1 | 9 | 2 | 14 | 26
percentage of participants | 100 [90.8 to 100.0] | 100 [20.7 to 100.0] | 100 [70.1 to 100.0] | 100 [34.2 to 100.0] | 92.9 [68.5 to 98.7] | 96.2 [81.1 to 99.3]

15. Secondary Outcome: Parts 1 & 2: Percentage of Participants With Sustained Virologic Response 24 Weeks After the Last Actual Dose of Study Drug (SVR24), Summarized by Formulation, Age and Weight Group, Across All Subjects, and Across All Subjects on the Adult Formulations
Description: SVR24 is defined as hepatitis C virus ribonucleic acid (HCV RNA) < lower limit of quantification (LLOQ) 24 weeks after the last actual dose of study drug.
Time Frame: 24 weeks after last dose of study drug (Week 36 or 48 depending on treatment duration)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Participants in Parts 1 and 2 of the Study: Participants in Parts 1 and 2 who were part of the ITT population (those who received at least one dose of study drug in Part 1 or Part 2)
Arm/Group | Participants in Parts 1 and 2 of the Study | Adult Tablet, 12-17 YR, ≥ 45 kg | Mini-tablet, 9-11 YR, 15 to 29 kg | Mini-tablet, 9-11 YR, 30 to 44 kg | Mini-tablet, 9-11 YR, ≥ 45 kg | Mini-tablet, 3-8 YR, 15 to 29 kg | Mini-tablet Total
Number analyzed (Participants) | 64 | 38 | 1 | 9 | 2 | 14 | 26
percentage of participants | 96.9 [89.3 to 99.1] | 100 [90.8 to 100.0] | 100.0 [20.7 to 100.0] | 88.9 [56.5 to 98.0] | 100.0 [34.2 to 100.0] | 92.9 [68.5 to 98.7] | 92.3 [75.9 to 97.9]

16. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization During Treatment by Formulation, Age and Weight Group, Across All Subjects, and Across All Subjects on the Adult Formulations
Description: Alanine aminotransferase (ALT) normalization during treatment is defined as ALT ≤ the upper limit of normal (ULN) at the final treatment visit for participants with ALT > ULN at baseline.
Time Frame: 12 or 24 weeks after starting study drug, depending on treatment duration
Population: Intention-to-treat population including participants whose alanine aminotransferase (ALT) levels were > the upper limit of normal at baseline and who had available on-treatment ALT data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Adult Tablet,12-17 YR, ≥ 45 kg, ALT Normalization: Participants age 12-17 years old with alanine aminotransferase > upper limit of normal at baseline who received the adult formulation and weighed ≥ 45 kg
- Mini-tablet, 9-11 YR, 15 to 29 kg, ALT Normalization: Participants age 9-11 years old with alanine aminotransferase > upper limit of normal at baseline who received the mini-tablet formulation and weighed 15 to 29 kg
- Mini-tablet, 9-11 YR, 30 to 44 kg, ALT Normalization: Participants age 9-11 years old with alanine aminotransferase > upper limit of normal at baseline who received the mini-tablet formulation and weighed 30 to 44 kg
- Mini-tablet, 3-8 YR, 15 to 29 kg, ALT Normalization: Participants age 3-8 years old with alanine aminotransferase > upper limit of normal at baseline who received the mini-tablet formulation and weighed 15 to 29 kg
- Mini-tablet Total, ALT Normalization: All participants with alanine aminotransferase > upper limit of normal at baseline who received the mini-tablet formulation
- Participants in Parts 1 and 2 of the Study, ALT Normalization: All participants with alanine aminotransferase > upper limit of normal at baseline
Arm/Group | Adult Tablet,12-17 YR, ≥ 45 kg, ALT Normalization | Mini-tablet, 9-11 YR, 15 to 29 kg, ALT Normalization | Mini-tablet, 9-11 YR, 30 to 44 kg, ALT Normalization | Mini-tablet, 3-8 YR, 15 to 29 kg, ALT Normalization | Mini-tablet Total, ALT Normalization | Participants in Parts 1 and 2 of the Study, ALT Normalization
Number analyzed (Participants) | 24 | 1 | 5 | 10 | 16 | 40
percentage of participants | 87.5 [69.0 to 95.7] | 100 [20.7 to 100.0] | 100 [56.6 to 100.0] | 80.0 [49.0 to 94.3] | 87.5 [64.0 to 96.5] | 87.5 [73.9 to 94.5]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 30 days after last dose, up to 37 weeks. SAEs and protocol-related nonserious AEs were collected from the time the subject signed consent.
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of study drug is administered until 30 days have elapsed following discontinuation of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Groups:
- Adult Tablet, 12-17 yr, Total: Participants age 12-17 years old who received at least one dose of the adult formulation
- Mini Tablet, Total: Participants who received at least one dose of the mini-tablet formulation
Arm/Group | Adult Tablet, 12-17 yr, Part 1 | Adult Tablet, 12-17 yr, Part 2 | Adult Tablet, 12-17 yr, Total | Mini Tablet, 9-11 yr, Part 1 | Mini Tablet, 3-8 yr, Part 1 | Mini Tablet, Total | All Participants, Total
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/26 | 0/38 | 0/12 | 0/14 | 0/26 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/26 | 0/38 | 1/12 | 0/14 | 1/26 | 1/64
Other Adverse Events (participants affected / at risk) | 11/12 | 17/26 | 28/38 | 12/12 | 9/14 | 21/26 | 49/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Tablet, 12-17 yr, Part 1 (N=12) | Adult Tablet, 12-17 yr, Part 2 (N=26) | Adult Tablet, 12-17 yr, Total (N=38) | Mini Tablet, 9-11 yr, Part 1 (N=12) | Mini Tablet, 3-8 yr, Part 1 (N=14) | Mini Tablet, Total (N=26) | All Participants, Total (N=64)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Tablet, 12-17 yr, Part 1 (N=12) | Adult Tablet, 12-17 yr, Part 2 (N=26) | Adult Tablet, 12-17 yr, Total (N=38) | Mini Tablet, 9-11 yr, Part 1 (N=12) | Mini Tablet, 3-8 yr, Part 1 (N=14) | Mini Tablet, Total (N=26) | All Participants, Total (N=64)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 4 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 7 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 5 (5) | 6 (6)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 5 (5) | 7 (7) | 5 (5) | 1 (1) | 6 (6) | 13 (13)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 3 (3) | 3 (4) | 2 (2) | 5 (6) | 8 (9)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (5) | 5 (6) | 2 (2) | 1 (2) | 3 (4) | 8 (10)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (3) | 4 (6) | 1 (1) | 3 (3) | 4 (4) | 8 (10)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram change (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 5 (5) | 8 (8) | 5 (6) | 2 (2) | 7 (8) | 15 (16)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Behavioural insomnia of childhood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sleep terror (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT02486406/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT02486406/SAP_001.pdf